CLINICAL TRIAL: NCT02836158
Title: Therapeutic Effects of R-IDARAM and Intrathecal Immunochemotherapy on Elderly Patients With Primary CNS Lymphoma
Brief Title: Therapeutic Effects of R-IDARAM and Intrathecal Immunochemotherapy on Elderly Patients With PCNSL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Doctor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NavyGHB-002
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-IDARAM plus intrathecal chemotherapy (Experimental): Patients will be treated with systemic R-IDARAM plus intrathecal immunochemotherapy
  Interventions: Drug: R-IDARAM plus intrathecal chemotherapy

INTERVENTIONS:
Drug: R-IDARAM plus intrathecal chemotherapy — R-IDARAM comprised of rituximab 375 mg/m2 (day 1), idarubicin 10 mg/m2(day 2); dexamethasone 100 mg/m2 (12 h.infusion in day 2, 3 and 4); cytarabine 1 g/m2 (1 h. infusion in day 2); methotrexate 1.5 g/m2 (6 h. infusion in day 4 with folinic acid rescue). Intrathecal Immunochemotherapy comprised of rituximab 20mg, MTX 15mg, dexamethasone 5mg and Ara-c 50mg once a week.
  Other Names: R-IDARAM plus intrathecal immuochemotherapy

SUMMARY:
This study suggests that R-IDARAM combined with intrathecal immunochemotherapy may be high effective in elderly patients with primary central nervous system lymphoma (PCNSL).

DETAILED DESCRIPTION:
The investigators will evaluate response rate, progression free survival (PFS), overall survival (OS), and toxicity in elderly patients with primary central nervous system lymphoma (PCNSL) after systemic and intrathecal immunochemotherapy with deferred radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically proven non-Hodgkin's lymphoma (NHL).

Exclusion Criteria:

* Involved sites other than the brain, meninges, CSF, or the eyes.
* Age less than 18 years or greater than 75 years.
* Inadequate bone marrow capacity (defined as neutrophils<1.5 ×10^9/L, platelets <100 ×10^9/L, and hemoglobin level< 8 g/dL).
* Known cause of immunosuppression (ie, HIV type I infection).
* Any previous malignancy.
* Creatinine clearance below 60 mL/min.
* Heart insufficiency (NYHA IIIB or IV).
* Uncontrolled infection.
* Noncompensated active pulmonary or liver disease.
* Previously treated for PCNSL, except by corticosteroids.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 year Overall survival
  3 year Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, M.D., Study Chair — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No